CLINICAL TRIAL: NCT03818633
Title: Effect of Elastic Abdominal Binder on Pain and Functional Recovery Following Gynecologic Cancer Surgery: a Randomized Controlled Trial
Brief Title: Elastic Abdominal Binder Following Gynecologic Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kittipat Charoenkwan, MD, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OBG-2560-05147
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic abdominal binder (Experimental)
  Interventions: Device: Elastic abdominal binder
- No binder (No Intervention)

INTERVENTIONS:
Device: Elastic abdominal binder — Each woman in the intervention group is fitted with an elastic abdominal binder at the time of procedure completion just before leaving the operating room. The binder is placed snuggly tight (keeping in mind patient's comfort) on top of the hospital gown with the incision positioned at the middle part of the binder. The patients are encouraged to wear binders at all time. However, periods of break from wearing the binder are allowed at their convenience.
  Arms: Elastic abdominal binder

SUMMARY:
Surgery is the primary treatment for gynecologic malignancies. The surgical approach provides opportunities for removal of the affected organs and complete assessment of extent of cancer spread. However, the procedures are often associated with significant morbidity. This is especially true with open laparotomy, the most frequently employed approach in developing countries. Delayed functional recovery influenced by pain and immobilization are important contributing factors for increased morbidity. Elastic abdominal binder, a wide elastic belt that is wore around the patient's abdomen to support surgical incision after surgery, has been employed by clinicians for pain relief, wound complications prevention, improved pulmonary function, and stabilization. Benefits of the abdominal binder use in this patient population have not been properly examined.

The aim of this study is to examine the effect of postoperative elastic abdominal binder use on recovery by comparing pain scores and mobility function (through the 6-minute walk test [6MWT]) in postoperative gynecologic cancer patients who use versus do not use the elastic abdominal binder to support incisional site.

ELIGIBILITY:
Inclusion Criteria:

* Women, diagnosed with gynecologic malignancies (carcinoma of the cervix, endometrium, and ovary), undergoing open abdominal surgery

Exclusion Criteria:

* Intraoperative accidental injury to urinary or gastrointestinal organs
* Postoperative admission to intensive care unit (ICU)
* Postoperative intraperitoneal drain placement
* Unable to understand and follow oral/written instructions
* Severe neuromuscular or circulatory disorders

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Daily average postoperative pain scores | An average of pain scores at 8:00 am and 4:00 pm, up to 7 days postoperation
  The participants are asked to rate postoperative pain according to 10-cm visual analog scales from '0' (no pain) to '10' (worst possible pain).
Six-minute walk test score change from baseline | One day before operation and postoperative day 3
  Six-minute walk test (6MWT)

SECONDARY OUTCOMES:
Quality of life: EuroQol Group's ED-5D-5L questionnaire | In the morning of postoperative day 3
  The EuroQol Group's ED-5D-5L questionnaire is employed. The health dimensions assessed include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each dimension, the participants are asked to indicate their health state related to that dimension as no problems (score '1'), slight problems (score '2'), moderate problems (score '3'), severe problems (score '4'), and extreme problems (score '5'). For this study, a score of 1-2 is considered "normal" while a scores of 3-5 is regarded as "problem". In addition, the participants are asked to rate their overall health status according to a visual analog scale EQ VAS with '0' corresponding to "the worst health imaginable" and '100' indicating "the best health imaginable".
Rate of postoperative complications | In the morning, up to 7 days postoperation
  The complications of interest include febrile morbidity, wound complication, bowel ileus

CONTACTS AND LOCATIONS:
Overall Officials: Kittipat Charoenkwan, MD, MSc, Principal Investigator — Chiang Mai University
Locations (1):
- Kittipat Charoenkwan, Chiang Mai, Thailand